CLINICAL TRIAL: NCT00672880
Title: The Use of Self-System Therapy to Alter Self-Discrepancies in Chronic Low Back Pain Patients
Brief Title: Self System Therapy and Chronic Low Back Pain Trial
Acronym: Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006455; NINDS Grant: RO 1NSO46422
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2015-03

CONDITIONS: Low Back Pain; Depression
Keywords: Chronic low back pain accompanied by depression
MeSH Terms: conditions — Low Back Pain; Depression | interventions — Educational Status; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Psychotherapy
  Interventions: Behavioral: Self-System Therapy
- 2 (Active Comparator): Spine Education
  Interventions: Behavioral: Education
- 3 (Placebo Comparator): Standard Care
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Self-System Therapy — 12 sessions of structured Self-System Therapy
  Arms: 1
Behavioral: Education — 12 sessions of spine and muscle education including life style changes and medical treatments.
  Arms: 2
Other: Standard Care — Study participants continue with their usual medical care, no changes.
  Arms: 3

SUMMARY:
This study is for people with chronic low back pain who may also be feeling discouraged, frustrated, or depressed. This study is testing a new therapy that is designed to specifically help these patients foster a better self-image. We hope this therapy will help them feel less discouraged and depressed and, possibly, even help reduce their stress enough that they may feel less pain.

DETAILED DESCRIPTION:
Patients with chronic low back pain cope with numerous life challenges, including the ability to work and decrements in physical and emotional well being. These changes impact the patients' abilities to pursue and achieve not only important personal and professional goals, but also make it difficult to maintain one's general standards of quality of daily life with personal tasks.

This study aims to address the feelings and attitudes associated with these shortfalls which frequently result in depression.

Eligible participants have been undergoing treatment for low back pain and have been identified as depressed. Study participants are randomized into one of three arms:

Self System Therapy-Patients receive 12 sessions (90 Min) one-on-one with a specialized treatment regimen designed to help patients foster a better self-image and re-evaluate their life's goals in light of their new physical limitations. Modifications in goal unavailability, goal activation, and goal accomplishments are key components in this therapy delivered by a therapist.

Low Back Pain Education-Patients receive 12 sessions (90 min) of detailed information about chronic low back pain, its causes and varied treatments, delivered by a research nurse.

Standard Care-Patients receive their routine medical care and serve as a treatment control group. They receive the same follow up evaluations as the other two groups.

Measures- Before each of the 4 evaluations, 30 day diaries are completed which measure daily pain coping, daily life events, daily mood and unpleasantness, and daily goal setting and accomplishments.

Patients are evaluated at 4 times, before treatment, after treatment, and at a 6 month and 12 month intervals. An interview version of the Selves Questionnaire is used to measure self-discrepancies. Pain behaviors are assessed by means of structured observation involving videotaping. Other outcome measures include questionnaires for depression, psychosocial disability, physical disability, and cognitive, affective, motivational, and physiological areas of depressive symptomology.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years and older
* Low back pain for minimum of 6 months
* DSM-IV diagnosis of major depressive disorder or dysthymia as determined by SCID interview, or meeting 18 or higher on Beck Depression Inventory.

Exclusion Criteria:

* Diagnosis of schizophrenia, bipolar, organic brain syndrome, substance abuse within past 5 years
* Hallucinations, delusions, or paranoid ideation
* Concurrent medical disorders that may cause depression or significantly affect function (epilepsy, endocrine disease, COPD, diabetes), or intellectual impairment based on clinical interview
* Inability to speak English; AND
* Patients with pending litigation or in the process of seeking disability benefits.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2003-10; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Depression levels | Post and 6 mo and 12 mo follow-up evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Francis Keefe, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States